CLINICAL TRIAL: NCT02487615
Title: Subclinical Atherosclerosis: Biomarkers of Early Disease
Brief Title: Genetical, Anthropometrical and Biochemical Factors Influencing High Risk Subclinical Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Adriana Bertolami, Adriana Bertolami, Instituto Dante Pazzanese de Cardiologia
Other Study IDs: 3852
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Primary Prevention
Keywords: Glycaemia; Subclinical Atherosclerosis; Carotid Doppler Ultrasound; Carotid Plaque; Intima Media Thickness; Ankle Brachial Index; Exercise Stress Test; Coronary Calcium Score; Insulinemia; Leptin; Inflammation; Resistin; Tumor Necrosis Factor alpha; Phospholipase A2, Group VII; Body Mass Index; Adipose Tissue Function; Single Gene Polymorphism
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Whole blood, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Subclinical atherosclerosis is the atherosclerotic process identified before clinical symptoms and thus it can be a useful marker of future cardiovascular events. It can be evaluated by many methods. This study included the diagnosis of subclincal atherosclerosis by four different methods: coronary calcium score, carotid doppler ultrasound to quantify intima media thickness and carotid plaques, exercise stress test and ankle brachial index. Clinical data, anthropometric measures (body mass index, abdominal circumference), markers of inflammation (high sensitive - C reactive protein, TNF alfa and Lipoprotein Associated Phospholipase A2), fat tissue function (leptin, resistin and adiponectin), glucose metabolism (fasting plasma glucose, glycated hemoglobin and insulin) and genetics markers of atherosclerotic process were evaluated as biomarkers of subclinical atherosclerosis in a uneventful population.

DETAILED DESCRIPTION:
This study cross-sectionally evaluated consecutive patients at the outpatient clinic of Dyslipidemia and of Hypertension and Nephrology Medical Sections of Dante Pazzanese Institute of Cardiology, a cardiologic tertiary hospital in São Paulo - Brazil. After they fulfilled inclusion criteria and signed an informed consent, a brief medical history and anthropometric data (abdominal circumference, height and weight for body mass index calculation) were collected. Within of a month after inclusion, all patients underwent blood sample collection for dosing fast plasma glucose and insulin and 2 hours after 75g of dextrose test glucose and insulin, fast serum triglycerides, total cholesterol, HDL cholesterol, creatinine, high sensitive c-reactive protein (hs-CRP), HbA1c, thyroid stimulating hormone (TSH), free thyroxin (fT4), creatine kinase, adiponectin, resistin, leptin, tumor necrosis factor alpha (TNF-α), lipoprotein associated phospholipase A2 (Lp-PLA2). Blood sample was also stored for DNA (rs2383206, rs10757274, rs10757278, rs1051931, rs16874954 and rs1799724) and RNA PLA2G7 (2-ΔCT), TNF-α (2-ΔCT), LEP (2-ΔCT), LEPR (2-ΔCT) extraction and analyses.

Subclinical atherosclerosis was evaluated by four methods: carotid doppler ultrasound, cardiac computed tomography, exercise stress test and ankle-brachial index (ABI). All above tests were performed at the same day.

Carotid Doppler ultrasound was performed by using high-resolution Vivid 7 ultrasound (GE, USA) and high-frequency linear transducer type 9 MHz with automated measurement. Carotid Intima media thickness (cIMT) was evaluated 1 cm distal of the posterior wall of the left and right common carotid arteries and the presence of atherosclerotic plaques in common, internal and external carotid arteries was assessed. Carotid plaque was defined by the presence of focal wall thickening at least 50% greater than that of the surrounding vessel wall, or as a focal region with IMT greater than 1.5 mm, which protrude into the lumen and that is distinct from the adjacent boundary.

Cardiac Computed Tomography was performed to determine coronary calcium score (CAC) and calcium distribution. Hepatic density was performed to evaluate the presence of hepatic steatosis with Aquilion apparatus (Toshiba Medical, Tochigi, Japan) with 64 rows of detectors. The acquisition of tomographic data was represented by images of average thickness (3 mm) and low intensity (50 milliamps, 120 kV) and coupled to the electrocardiogram. Calcium score was considered present when its density in the coronary artery was above 130 Housfield units (HU) for at least 3 continuous pixels (> 1 mm2) of the same coronary artery. Calcium score comprised the sum of individual scores of the left and right coronary arteries.

Exercise stress test was performed following under one of following protocols: Bruce, modified Bruce or Ellestad treadmill. The test was interrupted if maximum heart rate was reached or if clinical symptoms installed, including exhaustion. The exam was considered positive when there were: negative horizontal/descending deflection of ST segment measured at the J point ≥1 mm, pain suggestive of coronary artery disease, complex and sustained ventricular arrhythmias, plateau or drop in systolic blood pressure in effort and/or functional capacity lower than 5 METS.

ABI tests were performed with the patient in the supine position after resting for five minutes. Palpation of bilateral arterial pulses of pedial, posterior tibial, popliteal and brachial were performed. Measures of systolic pressures were made by a 5 MHz ultrasonography. The relationship between systolic and diastolic pressures of upper and lower limbs was used for calculating the ABI. The test was considered positive when at least one of the relationships was less than 0.9.

Personal and clinical characteristics of the patients will be described according to group using absolute and relative frequencies for qualitative characteristics and summary measures (mean, standard deviation, median, minimum and maximum) for quantitative characteristics. Distribution of the variables will be tested using Kolmogorov-Smirnov test. Comparative analyses for non-normal data will be performed using Kruskal-Wallis test and expressed as median (interquartile range). Normal data will be evaluated using analyses of variance (ANOVA) and expressed as mean ± standard deviation. To evaluate associations between categorical variables chi-square test and Fisher's Exact test will be used. Analysis of covariance (ANCOVA) adjusted for age and sex will be used to compare clinical and biochemical measures between groups (glucose, insulin, Homa-R, hs-PCR, HDL-c, triglycerides, LDL-c, HbA1c, TNF-α, leptin, 2 hours glucose and regular use of medication). Ordinal logistic regression will be used to evaluate subclinical atherosclerosis. A two-tailed P value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals free of clinical manifested arterial atherosclerotic disease

Exclusion Criteria:

* Uncontrolled hypothyroidism
* Use of hypoglycemic medications
* Liver failure
* Chronic kidney disease stage IV or V
* Heart failure NYHA stage III or IV
* HIV positive patients
* Withdrawal of informed consent

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive individuals attended at the outpatient clinic of Dyslipidemia and of Hypertension and Nephrology Medical Sections of Dante Pazzanese Institute of Cardiology, a cardiologic tertiary hospital in São Paulo - Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Carotid intima-media thickness (cIMT) | Four Weeks
  Subclinical atherosclerosis evaluation by quantifying intima media thickness by Doppler

SECONDARY OUTCOMES:
Coronary artery calcium score | Four weeks
  Subclinical atherosclerosis evaluation by Coronary Artery Calcium by CT
Brachial Ankle Index | Four weeks
  Subclinical atherosclerosis evaluation by brachial ankle index (BAI) by blood pressure measurement
Ischemia induced by exercise stress test | Four weeks
  Myocardial ischemia investigation by treadmill exercise test
Adiponectin, resistin, leptin, tumor necrosis factor alpha (TNF-α), lipoprotein associated phospholipase A2 (Lp-PLA2) | Four weeks
  Blood samples for Adiponectin, resistin, leptin, tumor necrosis factor alpha (TNF-α), lipoprotein associated phospholipase A2 (Lp-PLA2) dosing
Genotyping of DNA at the following rs2383206, rs10757274, rs10757278, rs1051931, rs16874954 and rs1799724 and RNA of PLA2G7 (2-ΔCT), TNF-α (2-ΔCT), LEP (2-ΔCT), LEPR (2-ΔCT) | Four weeks
  DNA and extraction from leukocytes

CONTACTS AND LOCATIONS:
Overall Officials: Andriana Bertolami, MD, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Andrei C Sposito, MD, PhD, Study Chair — University of Campinas, Brazil
Locations (2):
- Brazil (2):
  - State University Of Campinas, Campinas, São Paulo
  - Dante Pazzanese Institute of Cardiology, São Paulo, São Paulo